CLINICAL TRIAL: NCT01187316
Title: Massage and Transcutaneous Electrical Nerve Stimulation Therapies for Temporomandibular Disorders in Adolescents
Brief Title: Treatment of Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Responsible Party: Arnaldo de França Caldas Junior, University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-R6YV8
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2007-03

CONDITIONS: Temporomandibular Joint Disorders
Keywords: Facial Pain; Temporomandibular Joint Disorders; Transcutaneous Electric Nerve Stimulation; Adolescent
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain | interventions — Transcutaneous Electric Nerve Stimulation; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TENS (Experimental)
  Interventions: Device: Transcutaneous electrical nerve stimulation
- Massage therapy and muscle stretching (Active Comparator)
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — Sensors were positioned on anterior temporal and masseter muscles bilaterally, and the stimulation was used for 20 minutes at 150 Hz and 100 µs of pulse width; intensity was adjusted individually.
  Arms: TENS
Other: Physiotherapy — Massage and stretching of the anterior temporal and masseter muscle were performed by an experienced professional for 20 minutes.
  Arms: Massage therapy and muscle stretching

SUMMARY:
The aim of the present study was to carry out a pilot project comparing the effectiveness of two therapeutic approaches to temporomandibular disorders (TMDs) in adolescents. Eight female individuals diagnosed based on the Research Diagnosis Criteria for TMDs (RDC/TMD-axis 1)were randomly divided into two groups: 1) Massage therapy and muscle stretching (n=4); and 2) transcutaneous electrical nerve stimulation (TENS) (n=4). Regardless the treatment, ten sessions were held for each patient and two measurements (baseline and 10th session) were performed for the assessment of symptom evolution using a visual analog scale (VAS), maximum opening of the mouth (MOM) and pressure pain threshold (PPT). Statistical analysis wiil be carefully selected.

ELIGIBILITY:
Inclusion Criteria:

* Pain in orofacial area for at least 3 months
* Diagnosed at group 1 of RDC/TMD (myofascial pain with or without mouth opening limit)

Exclusion Criteria:

* Drug use for treatment of pain
* Functional limitations that would harm diagnosis

Ages: 14 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2007-04; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Pain | Two times a week
  The subjects was asked to mark the intensity of the pain on a 100mm line, which was numbered from 0 to 10, being "0" = no pain, and 10 = to the worst pain ever felt. The outcome of pain intensity was given as a number marked by the patient.

SECONDARY OUTCOMES:
Maximum mouth opening amplitude | Two times a week
  Subjects were asked to open their mouths as much as they could and the opening amplitude was measured using a digital caliper.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaldo F Caldas Junior, PhD, Principal Investigator — University of Pernambuco; Silvia D Benevides, Ms, Study Director — Federal University of Bahia; Mauricio Kosminsky, PhD, Study Chair — University of Pernambuco
Locations (2):
- Brazil (2):
  - Faculty of Dentistry of Pernambuco; Orofacial Control Center, Camaragibe, Pernambuco
  - Faculty of Dentistry of Pernambuco; Orofacial Control Center, Recife, Pernambuco

REFERENCES:
- [Background] List T, Wahlund K, Larsson B. Psychosocial functioning and dental factors in adolescents with temporomandibular disorders: a case-control study. J Orofac Pain. 2001 Summer;15(3):218-27. PMID 11575192
- [Background] Visscher CM, Lobbezoo F, Naeije M. Comparison of algometry and palpation in the recognition of temporomandibular disorder pain complaints. J Orofac Pain. 2004 Summer;18(3):214-9. PMID 15509000
- [Background] Rodrigues D, Siriani AO, Berzin F. Effect of conventional TENS on pain and electromyographic activity of masticatory muscles in TMD patients. Braz Oral Res. 2004 Oct-Dec;18(4):290-5. doi: 10.1590/s1806-83242004000400003. PMID 16089258
- [Background] Nilsson IM. Reliability, validity, incidence and impact of temporormandibular pain disorders in adolescents. Swed Dent J Suppl. 2007;(183):7-86. PMID 17506471